CLINICAL TRIAL: NCT01984567
Title: The Effects of Consumption of Vitamin E or Lipoic Acid on Serum Oxyphytosterol Concentrations in Subjects With Impaired Glucose Tolerance or Type II Diabetes
Brief Title: Vitamin E or Lipoic Acid on Serum Oxyphytosterol Concentrations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Jogchem Plat, Professor, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: NL40392.068.12 / METC 12-3-047
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Oxidative Stress
Keywords: Oxyphytosterols; Oxidative stress; Vitamin E; Lipoic acid
MeSH Terms: interventions — Vitamin E; Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin E (Experimental)
  Interventions: Dietary Supplement: Vitamin E
- Lipoic acid (Experimental)
  Interventions: Dietary Supplement: Lipoic acid
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Vitamin E — Daily consumption of vitamin E capsules, 3 capsules of 268 mg daily, in total daily consumption of 804 mg
  Arms: Vitamin E
Dietary Supplement: Lipoic acid — Daily consumption of lipoic acid capsules, 3 capsules of 200 mg daily, in total daily consumption of 600 mg
  Arms: Lipoic acid
Dietary Supplement: Control — Daily consumption of 3 placebo capsules
  Arms: Control

SUMMARY:
Background of the study:

We now know that plant sterols can oxidize, which results in the formation of oxyphytosterols. Animal studies have suggested that oxyphytosterols are atherogenic components, however this relation has not yet been studied in humans. In our previous study (METC 09-3-088) we have shown in healthy volunteers that serum oxyphytosterol concentrations are linked to oxidative stress status (i.e. we were able to identify high and low sterol oxidizers). From the literature is known that especially type II diabetics and IGT subjects are characterized by increased oxidative stress markers and reduced antioxidant capacity. For this reason we also want to evaluate the oxyphytosterol concentrations in this population. Moreover, we know propose to evaluate the effect of antioxidant supplementation, i.e. vitamin E or lipoic acid, on serum oxyphytosterol concentrations in type II diabetic patients. If possible to lower oxyphytosterol concentrations in these populations this is obviously beneficial in case oxyphytosterols turn out to be atherogenic. The major objective of the present study is to examine the effect of consuming vitamin E (804 mg) or lipoic acid (600 mg) for 4 weeks on fasting oxyphytosterol concentrations in subjects with impaired glucose tolerance or type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years
* Body Mass Index (BMI) between 20-35 kg/m2
* Mean serum total cholesterol <8.0 mmol/L
* Mean serum triacylglycerol <3.0 mmol/L
* Diagnosed with diabetes mellitus type 2 on a clinical basis or impaired glucose tolerance (defined as blood glucose >7.8 mmol/l and <11.0 mmol/L, two hours after ingesting 75 gram glucose in 150 ml water)

Exclusion Criteria:

* Unstable body weight (weight gain or loss > 3 kg in the past two months)
* Active cardiovascular diseases like congestive heart failure or recent (<6 months) event (acute myocardial infarction, cerebral vascular incident)
* Severe medical conditions that might interfere with the study such as epilepsy, asthma, chronic obstructive pulmonary disease, inflammatory bowel disease and rheumatoid arthritis
* Use of medication such as corticosteroids, diuretics or lipid lowering therapy
* Use of insulin therapy
* Abuse of drugs or alcohol (>21 units per week)
* Not willing to stop the consumption of vitamin supplements, containing lipoic acid and/or vitamin E, 1 month before the start of the study (wash-in period)
* Use of an investigational product within another biomedical study within the previous month
* Pregnant or breast-feeding women
* Current smoker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Plasma oxyphytosterol concentrations | Measured after 4 weeks intervention

SECONDARY OUTCOMES:
Serum lipoprotein concentrations | Measured after 4 weeks intervention
Markers reflecting oxidative stress | Measured after 4 weeks intervention
Markers reflecting antioxidant capacity | Measured after 4 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, Prof., Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands